CLINICAL TRIAL: NCT03383328
Title: Effect of Drop-less Surgery Compared to Topical NSAID Alone and Combination of Steroid and NSAID on Central Macular Thickness After Cataract Surgery, a Randomized Controlled Trial
Brief Title: Study for Optimizing Anti-inflammatory Prophylaxis
Acronym: SOAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Line Kessel (Other)
Responsible Party: Sponsor-Investigator, Line Kessel, Consultant ophthalmologist, Associate Professor, MD, Ph.D., FEBO, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SOAP1
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Cystoid Macular Edema; Irvine-Gass Syndrome
Keywords: Cataract; Cataract Surgery
MeSH Terms: conditions — Macular Edema; Cataract | interventions — Anti-Inflammatory Agents, Non-Steroidal; Prednisolone; Postoperative Period; SOXB2 Transcription Factors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- NSAID + prednisolone, preoperative (Active Comparator): Combination of NSAID- and prednisolone eye drops. Treatment is initiated 3 days prior to surgery and administered 3 times pr. day for 3 weeks.
  Ketorolactrometamol 5 mg/ml, eye drops, 1 drop 3 times pr. day Prednisolone acetate 1% w/v, eye drops, 1 drop 3 times pr. day
  Interventions: Drug: NSAID + prednisolone, preoperative
- NSAID + prednisolone, postoperative (Active Comparator): Combination of NSAID- and prednisolone eye drops. Treatment is initiated on the day of surgery and administered 3 times pr. day for 3 weeks.
  Ketorolactrometamol 5 mg/ml, eye drops, 1 drop 3 times pr. day Prednisolone acetate 1% w/v, eye drops, 1 drop 3 times pr. day
  Interventions: Drug: NSAID + prednisolone, postoperative
- NSAID, preoperative (Experimental): NSAID eye drops as monotherapy. Treatment is initiated 3 days prior to surgery and administered 3 times pr. day for 3 weeks.
  Ketorolactrometamol 5 mg/ml, eye drops, 1 drop 3 times pr. day
  Interventions: Drug: NSAID, preoperative
- NSAID, postoperative (Experimental): NSAID eye drops as monotherapy. Treatment is initiated on the day of surgery and administered 3 times pr. day for 3 weeks.
  Ketorolactrometamol 5 mg/ml, eye drops, 1 drop 3 times pr. day
  Interventions: Drug: NSAID, postoperative
- Drop-less surgery (Experimental): A depot of dexamethasone is administered subtenonally during surgery.
  Dexamethason Krka 4 mg/ml solution for injection/infusion. 0,5 ml equivalent to 2 mg of dexamethasone is administered once.
  Interventions: Drug: Drop-less surgery

INTERVENTIONS:
Drug: NSAID + prednisolone, preoperative — Ketorolactrometamol 5 mg/ml and prednisolone acetate 1% w/v eye drops are administered 3 times pr. day, starting 3 days prior to surgery and until 3 weeks after surgery.
  Other Names: Group a1
  Arms: NSAID + prednisolone, preoperative
Drug: NSAID + prednisolone, postoperative — Ketorolactrometamol 5 mg/ml and prednisolone acetate 1% w/v eye drops are administered 3 times pr. day, starting on the day of surgery and until 3 weeks after surgery.
  Other Names: Group a2
  Arms: NSAID + prednisolone, postoperative
Drug: NSAID, preoperative — Ketorolactrometamol 5 mg/ml eye drops are administered 3 times pr. day, starting 3 days prior to surgery and until 3 weeks after surgery.
  Other Names: Group b1
  Arms: NSAID, preoperative
Drug: NSAID, postoperative — Ketorolactrometamol 5 mg/ml eye drops are administered 3 times pr. day, starting on the day of surgery and until 3 weeks after surgery.
  Other Names: Group b2
  Arms: NSAID, postoperative
Drug: Drop-less surgery — A depot of 0.5 ml Dexamethason Krka 4 mg/ml solution for injection/infusion is administered during cataract surgery.
  Other Names: Group c
  Arms: Drop-less surgery

SUMMARY:
The purpose of this study is to investigate which anti-inflammatory treatment is best at preventing postoperative inflammation following cataract surgery. We want to compare topical prophylaxis with NSAID eye drops to topical prophylaxis with a combination of NSAID and prednisolone. We also want to compare topical prophylaxis with eye drops to drop-less surgery where the anti-inflammatory drug is administered to the subtenonal space at the conclusion of the surgical procedure. In addition, we want to investigate if topical anti-inflammatory prophylaxis should be initiated preoperatively or postoperatively. The primary outcome is change in central macular thickness, measured by optical coherence tomography, 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age-related cataracts
* Older than 18 years
* Women must be postmenopausal. Women are asked if they have menstruated within the preceding 12 months.
* Capacity to consent
* Scheduled to undergo cataract surgery at the ophthalmic department at Rigshospitalet-Glostrup, Denmark
* The surgeon must be experienced, defined by a minimum of 1000 cataract extractions completed
* Only 1 eye can be included for each participant, but there are no restrictions as to whether it is the eye that undergoes surgery first or last. If both eyes of a participant are eligible, it will be decided by randomization which eye to be included in the study
* Informed consent to participation

Exclusion Criteria:

* Known allergy to any of the contents of the pharmaceuticals (active and in-active ingredients) used in the study
* Medical history of epiretinal membrane, retinal vein occlusion, retinal detachment, uveitis, glaucoma, diabetes mellitus, exudative age-related macular degeneration (AMD) or AMD with geographical atrophy
* Significant complications to surgery such as posterior capsule rupture/vitreous loss, choroidal hemorrhage, and dislocated lens material
* Pregnancy
* Fertile women, i.e. women who are not menopausal.
* Women who breastfeed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | 3 months
  Change in central macular thickness (CMT) measured by optical coherence tomography 3 months after cataract surgery.

SECONDARY OUTCOMES:
Best corrected visual acuity | 3 days, 3 weeks and 3 months
  Postoperative best corrected visual acuity in logarithm to the minimal angle of resolution (logMAR)
Intraocular pressure | 3 days, 3 weeks and 3 months
  Change in intraocular pressure
Optical nerve damage | 3 weeks and 3 months
  Optical nerve damage, assessed by measuring retinal nerve fiber layer (RNFL) by peripapillary optical coherence tomography (OCT)
Flare and number of cells | 3 days
  Flare and number of cells measured by laser flare-cell photometry
Subjective patient tolerance | 3 days and 3 weeks
  Subjective patient tolerance of prophylactic treatment measured on a 4-point analog scale, where 0 = no discomfort, 1 = mild discomfort, 2 = moderate discomfort and 3 = severe discomfort.
Patient related outcome measures | 3 months
  Visual function questionnaires are filled out at baseline and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Line Kessel, MD, Ph.D., Principal Investigator — Dpt. of Ophthalmology, Rigshospitalet-Glostrup
Locations (1):
- Department of Ophthalmology, Glostrup Municipality, Capital Region, Denmark

REFERENCES:
- [Derived] Erichsen JH, Holm LM, Forslund Jacobsen M, Forman JL, Kessel L. Prednisolone and Ketorolac vs Ketorolac Monotherapy or Sub-Tenon Prophylaxis for Macular Thickening in Cataract Surgery: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Oct 1;139(10):1062-1070. doi: 10.1001/jamaophthalmol.2021.2976. PMID 34383010
- [Derived] Erichsen JH, Forman JL, Holm LM, Kessel L. Effect of anti-inflammatory regimen on early postoperative inflammation after cataract surgery. J Cataract Refract Surg. 2021 Mar 1;47(3):323-330. doi: 10.1097/j.jcrs.0000000000000455. PMID 33086290